CLINICAL TRIAL: NCT07189286
Title: Preserving Ability Through Virtual Exercise (PAVE): An Intervention to Increase the Physical Activity of Hospitalized Older Adults
Brief Title: Preserving Ability Through Virtual Exercise (PAVE)
Acronym: PAVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH); The Claude D. Pepper Older Americans Independence Centers (Other)
Responsible Party: Principal Investigator, Brittany Burch, Assistant Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1K01AG090761-01A1 (NIH); 1K01AG090761-01A1 (NIH)
Record Dates: First submitted 2025-09-09; First posted 2025-09-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Feasibility Studies

STUDY DESIGN:
Intervention Model Description: This proposed study, Preserving Ability through Virtual Exercise (PAVE), will be a quasi-experimental trial among hospitalized older adults. We plan to recruit the 140 participants from one medical floor, with 70 in the intervention group and 70 in the control group. Recruitment will occur in blocks. First, during the pilot phase, we will recruit 10 intervention participants and then 10 control participants, followed by a temporary pause in recruitment to assess feasibility data and identify any needed protocol refinements. If any refinements are needed, we will submit an IRB modification. Next, we will resume recruitment of 30 intervention and then 30 control participants, followed by 30 intervention and then 30 control participants. Randomizing participants within unit is not feasible because control participants could be exposed to the intervention by observing or interacting with intervention participants (e.g., roommates performing the intervention.
Masking Description: Participants will not be blinded to the behavioral intervention they are receiving. However, we have designed this study with sequential (blocked) recruitment to minimize bias due to awareness of another group, such as a control group participant being roommates with a PAVE participant as they perform virtual reality physical activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAVE intervention (Experimental): PAVE participants will be trained to use the virtual reality headset and perform virtual reality physical activity throughout their hospital stay.
  Interventions: Behavioral: PAVE intervention
- Education control (Active Comparator): Education control will receive physical activity education using the NIH "Get Fit for Life" booklet.
  Interventions: Behavioral: Education control

INTERVENTIONS:
Behavioral: PAVE intervention — The commercial virtual reality app that will be used for the intervention, Supernatural, provides participants a trainer as they use their arms and legs (e.g., seated knee strikes) to smash targets to 500+ musical tracks. In this manner, this study employs fun as a motivator for exercise commencement and adherence while hospitalized. The research assistant will implement the intervention using the three-step approach including: (1) patient mobility screen, (2) orientation to the technology and intervention, and (3) ongoing assessment, adaptation, and motivation.
  Other Names: virtual reality physical activity
  Arms: PAVE intervention
Behavioral: Education control — Education control participants will receive and physical activity education using the NIH "Get Fit for Life" booklet.
  Arms: Education control

SUMMARY:
Each day in the hospital leads to functional decline and loss of muscle mass, which older adults can find difficult or impossible to restore in the post-acute period. The overall objective of this proposed project is to explore the feasibility and preliminary efficacy of a virtual reality physical activity intervention at helping older adults engage in physical activity and maintain physical function and mental health during their hospital stay. As virtual reality technology becomes more affordable and ubiquitously available across the world, this study will demonstrate how this technology could be leveraged to maintain the function of older adults in the hospital.

DETAILED DESCRIPTION:
Older adults (≥60 years) experience multi-level barriers to physical activity when hospitalized. Patient level barriers to physical activity when hospitalized include tethers (e.g., foley catheters, intravenous infusions), symptoms of their acute illness (e.g., pain, fatigue), low self-efficacy to perform physical activity, and a perception that they should remain on bedrest when hospitalized. Interpersonal barriers to physical activity, highlighted during this post pandemic environment, include staffing shortages and increased patient acuity, which can force nurses to prioritize other critical tasks over the physical activity of their patients. Environmental barriers to physical activity include bed alarms and a hospital climate that is hyper focused on the incorrect assumption that physical activity increases fall risk among hospitalized older adults.

This lack of physical activity in the hospital generates major personal and societal costs. Each day a patient spends in the hospital increases their risk of functional decline and loss of muscle mass, which older adults can find difficult or impossible to restore in the post-acute period. Hospital associated deconditioning increases the length of hospital stays, and increases the susceptibility of patients to delirium, falls, and re-admission. Such complications ultimately increase health care costs. Therefore, there is a significant unmet need to identify strategies to increase older patients' physical activity while minimizing staff burden.

The overall objective of this proposed project is to explore the feasibility and preliminary efficacy of a virtual reality physical activity intervention to engage older adults in physical activity and maintain physical function and mental health during their hospital stay. This quasi-experimental study has two aims.

Primary) Aim 1: Using the NIH Behavior Change consortium guidelines, the Acceptability/Appropriateness of Intervention Measure, the Simulator Sickness Questionnaire, and semi-structured individual interviews, determine the feasibility of a virtual reality intervention among hospitalized older adults.

Aim 2: Test the preliminary efficacy of the PAVE intervention on 1) time spent in physical activity during the hospital stay, 2) maintenance of physical function, and 3) maintenance of mental health, compared to the education only control group.

Hypothesis 2.1. Patients exposed to the PAVE intervention will demonstrate more time spent in physical activity (MotionWatch, Modified Physical Activity Vital Sign) during their hospital stay, when compared to those exposed to the education control, controlling for appropriate covariates.

Hypothesis 2.2. Patients exposed to the PAVE intervention will better maintain their physical function throughout their hospital stay (Barthel Index, UMove), when compared to those exposed to the education control, controlling for appropriate covariates.

Hypothesis 2.3. Patients exposed to the PAVE intervention will better maintain their mental health throughout their hospital stay (Hospital Anxiety and Depression Scale, Brief Reslience Scale), when compared to those exposed to the education control, controlling for appropriate covariates.

ELIGIBILITY:
Inclusion Criteria:

1. in the last 48 hours, they were admitted to the medical floor that is the setting of the study,
2. are 60 years or older,
3. their bedside nurse approves their physical activity participation in this study

Exclusion Criteria:

1. they are unable to pass the Evaluation to Sign Consent Measure,
2. they score 23 or lower on the Montreal Cognitive Assessment,
3. they have a diagnosis that could be worsened through virtual reality exercise (e.g., nausea, syncope, vertigo, upper extremity fractures/sprain/strain),
4. they have an attached medical device that decreases the safety of physical activity such as a nasogastric tube or continuous fluids running through a PICC line that cannot be paused, or
5. they are unable to follow commands or move their extremities against gravity during the UMove Mobility Assessment
6. they are unable to wear the virtual reality headset
7. they received the education control intervention or PAVE intervention during a prior admission

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Acceptability of Intervention Measure | measured at discharge or 7 days post baseline, whichever occurs first
  Scores range from 4-20, with higher scores indicating greater acceptability of intervention
Feasibility: Appropriateness of Intervention Measure | measured at discharge or 7 days post baseline, whichever occurs first
  Scores range from 4-20, with higher scores indicating greater appropriateness of intervention
Feasibility: Simulator Sickness Questionnaire | measured following PAVE participants' first virtual reality session only; baseline only
  Scores range from 0 to 48, with higher score indicating more simulator sickness.
Feasibility: Qualitative Interviews | measured at discharge or 7 days post baseline, whichever occurs first (PAVE participants only)
  The interviews will include the following four questions: (1) "What did you like best about the virtual reality physical activity intervention?", (2) "What did you like least about the virtual reality physical activity intervention?", (3) "How, if at all, did participating in the virtual reality exercises affect the way you coped with challenges during your hospital stay?" and (4) "How could this virtual reality physical activity intervention be improved?"

SECONDARY OUTCOMES:
Physical Activity | At baseline enrollment, we will apply the MotionWatch8 to participants' wrists. At discharge, or 7 days after baseline, whichever occurs first, we will remove the MotionWatch8.
  The MotionWatch8 is a lightweight, wrist-worn activity monitoring device with a battery that lasts approximately one month. The MotionWatch8 contains a valid and reliable accelerometer, which records physical movement of the wrist providing a close correlation to whole body movement (1-minute epochs, 50 Hz). We will quantify counts of activity into sedentary, light, moderate, and vigorous activity per day (as defined by Landry and colleagues, 2015, Front Aging Neurosci).
Physical Activity: Modified Physical Activity Vital Sign | Measured at baseline and discharge, or 7 days post baseline, whichever occurs first
  The modified Physical Activity Vital sign measures patients' self-report participation in physical activity. The 6 items gather if (yes/no) activity was performed, duration (in minutes), and intensity (ordinal 0-10, with higher scores indicating higher intensity) for movement and strength based activities within the last 24 hours.
Physical Function: Barthel Index | Measured at baseline and discharge, or 7 days post baseline, whichever occurs first
  Barthel Index. Scores range from 0-100, with higher scores indicating greater independence.
Physical Function: UMove Mobility Screen | Measured at baseline and discharge, or 7 days post baseline, whichever occurs first
  The UMove Mobility Scale is a clinical screening tool designed to help healthcare providers assess a patient's functional mobility and determine safe strategies for out-of-bed movement and ambulation. While there is no fixed numerical range, patients are categorized into mobility levels 1-5.
Mental Health: Hospital Anxiety and Depression Scale | Measured at baseline and discharge, or 7 days post baseline, whichever occurs first
  Hospital Anxiety and Depression Scale: Scores range from 0-21, with higher score indicating greater mental illness.
Brief Resilience Scale | Measured at baseline and discharge, or 7 days post baseline, whichever occurs first
  The Brief Resilience Scale is a 6-item ordinal scale that measures resilience. Greater scores indicate higher resilience. Scores range from 6-30, with higher scores indicating higher resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Burch, PhD, MSN, RN, Principal Investigator — University of Maryland Baltiomre
Locations (1):
- UMMC Midtown Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
During informed consent, study participants will be asked to consent to de-identified quantitative data sharing upon recommendations of the local IRB. We will share all collected quantitative data in a de-identified format (age, comorbidities, feasibility, physical activity, physical function, and mental health), removing all personal identifying information. All direct participant identifiers (e.g., name, date of birth) will be removed from data prior to sharing. Users of the generalist repository that will store this study's data, Zenodo, must agree to the Terms and Conditions of Zenodo, and agree not to share or redistribute the data. We will not share the transcripts from the qualitative individual interviews.
Supporting Information: Study Protocol, Analytic Code
Time Frame: We will actively disseminate the findings of the proposed project via standard peer review mechanisms including the submission of abstracts for poster and podium presentations at scientific meetings and the publication of peer reviewed articles.
  Data will be stored and maintained on University of Maryland's HIPAA-compliant servers. We will make all de-identified quantitative data publicly available upon publication of the work related to this proposed project, or the end of the project period, whichever comes first. This de-identified data will remain available indefinitely on Zenodo, a generalist repository supported by the NIH.
Access Criteria: Users of the generalist repository that will store this study's data, Zenodo, can access the individual quantitative data collected from this study, including information related to age, comorbidities, feasibility, physical activity, physical function, and mental health. All direct participant identifiers (e.g., name, date of birth) will be removed from data prior to sharing. We will not share the transcripts from the qualitative individual interviews.